CLINICAL TRIAL: NCT05448898
Title: The Efficacy of Traditional Chinese Medicine in Olfactory Dysfunction: A Randomized Controlled Trial
Brief Title: The Efficacy of Traditional Chinese Medicine in Olfactory Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ODCT2002-6
Record Dates: First submitted 2022-07-04; First posted 2022-07-08 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Olfactory Disorder
Keywords: Olfactory Function
MeSH Terms: interventions — Olfactory Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Chinese Medicine with olfactory training (Experimental): Traditional Chinese Medicine therapy:
  Oral Traditional Chinese Medicine CU Xiu Tang once a day for at least 3 months
  Olfactory training:
  repeat and deliberate sniffing of a set of odorants for 20 seconds each at least twice a day for at least 3 months
  Interventions: Drug: Traditional Chinese Medicine CU Xiu Tang; Other: Olfactory Training
- Olfactory training (Experimental): repeat and deliberate sniffing of a set of odorants for 20 seconds each at least twice a day for at least 3 months
  Interventions: Other: Olfactory Training

INTERVENTIONS:
Drug: Traditional Chinese Medicine CU Xiu Tang — Oral Traditional Chinese Medicine CU Xiu Tang once a day and repeat and deliberate sniffing of a set of odorants for 20 seconds each at least twice a day for at least 3 months
  Other Names: Olfactory Training
  Arms: Traditional Chinese Medicine with olfactory training
Other: Olfactory Training — repeat and deliberate sniffing of a set of odorants for 20 seconds each at least twice a day for at least 3 months

SUMMARY:
Studies have demonstrated that patients with olfactory dysfunction could improve the olfactory function after olfactory training. But the efficacy of Traditional Chinese Medicine is unknown.The purpose of this study is to evaluate its efficacy in olfactory dysfunction.

DETAILED DESCRIPTION:
A recent meta-analysis found significant positive effects of olfactory training on the individual subcomponents of odor threshold, discrimination, identification, and the composite TDI score. In addition to the evidenced improvement in olfactory function after olfactory training, this form of treatment carries very little risk of adverse effects, is cheap, and can be administered by the patient. For these collective reasons, olfactory training is an attractive treatment modality. Chinese experts consensus on diagnosis and treatment of olfactory dysfunction in 2017 shown that some evidences proved that Traditional Chinese Medicine treatment would benefit olfactory dysfunction but the evidences is not adequate. Until now, the efficacy of Traditional Chinese Medicine is controversial. This study investigate the efficacy and the safety of Traditional Chinese Medicine and olfactory training as a treatment for patients with olfactory dysfunction.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of Olfactory dysfunction;
2. 18 ≤ age ≤ 55 years old;
3. No active infection, such as uncontrolled pneumonia;
4. Women with reproductive potential and sexually active men agree to use acceptable and effective contraceptive methods.

Exclusion Criteria:

1. Refuse to sign informed consent;
2. With other diseases that affect the result, such as severe hepatic and renal dysfunction and the investigators believes will interfere with the treatment;
3. Pregnant or lactating women;
4. Without personal freedom and independent civil capacity;
5. Enrolled in other intervention clinical trials;
6. Autoimmune diseases;
7. Other situations that the investigators think are not suitable for the trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 278 (Estimated)
Dates: Start 2022-07-15 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Olfactory function test result | 3 months
  Olfactory tests combination of odor threshold (T), odor discrimination (D), and odor identification (I). The minimum values is 0, the maximum values of odor threshold (T), discrimination (D), and identification (I) is 16, the sum of the scores is TDI, which is between 0 to 48, the higher scores mean a better outcome.

SECONDARY OUTCOMES:
Odor threshold (T), Odor Discrimination (D), Odor Identification (I) | 3 months
  The scale of odor threshold (T), discrimination (D), and identification (I).The minimum values is 0, the maximum values of odor threshold (T), discrimination (D), and identification (I) is 16, the higher scores mean a better outcome.
the Visual Analogue Scale(VAS) of Olfactory Function | 3 months
  Participants should value their olfactory function by use the Visual Analogue Scale#VAS), the minimum values is 0, the maximum values is 10, the higher scores mean a better outcome.

OTHER OUTCOMES:
Questionnaire of Olfactory Disorders | 3 months
  every patients should answer the Questionnaire of Olfactory Disorders and record the results. The answers should be agreed, Partially agreed and disagreed.

CONTACTS AND LOCATIONS:
Overall Officials: Hongmeng Yu, Dr, Principal Investigator — Eye & ENT Hospital, Fudan University; YanQing Li, Dr, Principal Investigator — Eye & ENT Hospital, Fudan University
Locations (1):
- Eye & ENT Hospital, Shanghai, Shanghai Municipality, China